CLINICAL TRIAL: NCT03161860
Title: Effect of Personalised Citizen Assistance for Social Participation (APIC) on Older Adults' Health and Social Participation: a Pragmatic Multicentre Randomised Controlled Trial (RCT)
Brief Title: Effect of Personalised Citizen Assistance for Social Participation(APIC) on Older Adults Health and Social Participation
Acronym: APIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mélanie Levasseur (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Mélanie Levasseur, Research Professor, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MP-31-2018-2424
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Community-dwelling Older Adults
Keywords: Program evaluation; Cost-effectiveness; Community participation; empowerment
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the type of intervention, coordinators, volunteers and participants will not be blinded to the interventions. However, they will not be informed about the study hypotheses. Research assistants and the statistician responsible for the analysis will be blinded to the intervention until completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalised citizen assistance (Experimental): The experimental group will receive the Personalised citizen assistance for social participation (APIC), i.e. weekly 3-hour personalised stimulation sessions by a trained volunteer over 12 months. Sessions will encourage empowerment, gradual mobilisation of personal and environmental resources, and community integration.
  Interventions: Behavioral: Personalised citizen assistance for social participation(APIC)
- Control group (No Intervention): The control group will receive the publicly-funded universal healthcare services available to all Quebecers.

INTERVENTIONS:
Behavioral: Personalised citizen assistance for social participation(APIC) — The APIC involves a non-professional attendant who, after 2 to 5 days of training, provides a two to three-hour stimulation session each week over a six to eighteen-month period targeting significant social and leisure activities that are otherwise difficult for older adults to accomplish.
  Arms: Personalised citizen assistance

SUMMARY:
Global aging and the growing burden of chronic diseases represent a challenge. Innovative interventions acting upon health determinants, like social participation, are required. Social participation, defined as the involvement of a person in activities that provide interactions with others in the community is critical to promote health and prevent disabilities. Many older adults do not have equitable opportunities to achieve full social participation, and interventions under-empower their personal and environmental resources and only reach a minority. To optimize current practices, the Personalised citizen assistance for social participation (APIC), an intervention demonstrated as being feasible and having positive impacts, needs further evaluation.

The first aim of this study is evaluate the impacts of the APIC on older adults' health, social participation, life satisfaction and healthcare services utilisation. The second aim is to evaluate the cost-effectiveness of the intervention. In parallel, the implementation of the APIC, including factors facilitating and impeding it, will be documented.

Concerning the first two objectives, two hypotheses are formulated: 1) the APIC will prevent a decline in older women's and men's health, social participation and life satisfaction, and reduce their use of healthcare services, and 2) the APIC will be associated with lower costs, from older adults', healthcare system and societal perspectives, including healthcare expenditures.

ELIGIBILITY:
Inclusion Criteria:

1. be aged 65 or older,
2. live at home or in seniors' residences,
3. be restricted in at least one instrumental activity of daily living (e.g. house cleaning, shopping), and
4. have a good understanding of French or English.

Exclusion Criteria:

* Moderate to severe cognitive impairments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
v2 of the 36-Item Short-Form Health Survey (SF-36) (''change'' is is being assessed) | Baseline, 12, 18, 24 months
  Physical and mental health

SECONDARY OUTCOMES:
Social participation scale | Baseline, 12, 18, 24 months
  Social participation
Life Satisfaction Index-Z | Baseline, 12, 18, 24 months
  Life Satisfaction
Use of healthcare services-Standardized questionnaire | every two months over a 2-year period
  Use of healthcare services

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Levasseur, Principal Investigator — Université de Sherbrooke; Research centre on aging
Locations (6):
- Canada (6):
  - Centre d'action bénévole Drummond, Drummondville, Quebec
  - Centre d'action bénévole Bellechasse-Lévis-Lotbinière, Lévis, Quebec
  - Service d'aide et de référencement Anjou (SARA-Anjou), Montreal, Quebec
  - Carrefour communautaire Montrose, Montreal, Quebec
  - Centre ABC, Montreal, Quebec
  - Accorderie de Sherbrooke, coopérative de solidarité, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Levasseur M, Chaintre-Prieur A, Dubois MF, Maisonneuve C, Filiatrault J, Vassiliadis HM. Strengths, challenges, and strategies for implementing pragmatic multicenter randomized controlled trials (RCTs): example of the Personalized Citizen Assistance for Social Participation (APIC) trial. Trials. 2024 Jun 27;25(1):415. doi: 10.1186/s13063-024-08248-w. PMID 38937798
- [Derived] Levasseur M, Dubois MF, Filliatrault J, Vasiliadis HM, Lacasse-Bedard J, Tourigny A, Levert MJ, Gabaude C, Lefebvre H, Berger V, Eymard C. Effect of personalised citizen assistance for social participation (APIC) on older adults' health and social participation: study protocol for a pragmatic multicentre randomised controlled trial (RCT). BMJ Open. 2018 Mar 31;8(3):e018676. doi: 10.1136/bmjopen-2017-018676. PMID 29605819